CLINICAL TRIAL: NCT04835467
Title: First-In-Human Intracoronary Dual-modal Optical Coherence Tomography and Fluorescence Lifetime Imaging (OCT-FLIM) In Patients Undergoing Percutaneous Coronary Intervention
Brief Title: First-In-Human Intracoronary OCT-FLIm In Patients Undergoing PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Jin Won Kim, Jin Won Kim, MD, PhD, Korea University Guro Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SRFC-IT1501-05
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Atherosclerosis Coronary Artery With Angina Pectoris; Atheroscleroses, Coronary; Atherosclerotic Plaque; Thin-cap fIbroatheroma; Atherosclerosis
Keywords: Fluorescence lifetime imaging; High-risk coronary plaque; Optical coherence tomography; Intravascular imaging; Biochemical imaging
MeSH Terms: conditions — Coronary Artery Disease; Plaque, Atherosclerotic; Atherosclerosis

STUDY DESIGN:
Intervention Model Description: Single group patient enrollment and scheduled 6-month follow-up assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intracoronary imaging (Experimental): Intracoronary imaging during PCI
  Interventions: Device: Dual-modal OCT-FLIm

INTERVENTIONS:
Device: Dual-modal OCT-FLIm — Intracoronary imaging using dual-modal OCT-FLIm catheter

SUMMARY:
Patients will undergo intracoronary imaging using combined optical coherence tomography-fluorescence lifetime imaging (OCT-FLIm) during percutaneous coronary intervention, and the obtained imaging data will be used to assess the efficacy of this dual-modal catheter imaging strategy in characterizing high-risk plaque.

DETAILED DESCRIPTION:
Fluorescence lifetime imaging (FLIm) is a novel imaging approach allowing label-free biochemical characterization of atherosclerotic plaque. A combined optical coherence tomography (OCT) and FLIm that can provide a simultaneous structural and biochemical assessment of atheroma has been constructed successfully. This study sought to investigate whether the dual-modal intravascular OCT-FLIm is able to characterize high-risk plaques in patients undergoing percutaneous coronary intervention.

Forty patients with multivessel coronary artery disease, who had at least one obstructive lesion (>70% diameter stenosis) that is considered suitable for PCI, will be included in the study. Culprit and mildly stenotic non-culprit plaques will be imaged using OCT-FLIm catheter.

Six-month follow-up assessment is systematically scheduled in all patients to assess temporal changes in FLIm signatures according to treatment strategies (medical therapy, interventional therapy etc).

ELIGIBILITY:
Inclusion Criteria:

* Age: greater than 20, less than 80
* Patients with significant coronary artery disease (diameter stenosis >70%) requiring coronary revascularization
* Reference vessel diameter: between 2.5 and 4.0 mm
* Obtained informed consent from voluntary participants before study enrollment

Exclusion Criteria:

* Complex coronary lesion (ostial lesion, unprotected left main lesion, chronic total occlusion, grafted vessels, etc)
* Reference vessel diameter: less than 2.5 mm, greater than 4.0 mm
* Coronary lesion with heavy calcification
* Hemodynamic instability during coronary intervention
* Contraindication to antithrombotic therapy
* Chronic renal insufficiency (Serum creatinine >2.0mg/dL)
* Severe liver dysfunction (AST/ALT > 5 times of upper normal limit)
* Pregnancy or potential pregnancy
* Life expectancy less than 1 year
* Patient refused to sign the informed consent at enrollment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Fluorescence lifetime measurement of plaque inflammation in the target/culprit or non-target/non-culprit lesion (nanosecond) | day 1
  Difference in fluorescence lifetime measurement reflecting plaque inflammation according to pre-specified plaque subtypes

SECONDARY OUTCOMES:
Fluorescence lifetime measurement of healed plaque in the target/culprit or non-target/non-culprit lesion (nanosecond) | day 1
  Difference in fluorescence lifetime measurement reflecting healed property according to pre-specified plaque subtypes
Fluorescence lifetime measurement of calcification in the target/culprit or non-target/non-culprit lesion (nanosecond) | day 1
  Difference in fluorescence lifetime measurement reflecting superficial calficiation according to pre-specified plaque subtypes

OTHER OUTCOMES:
6-month temporal changes in FLIm measurement of plaque inflammation in the target/culprit or non-target/non-culprit lesion (nanosecond) | 6 month
  6-month changes in inflammatory FLIm measurement
6-month temporal changes in FLIm measurement of healed plaque phenotype in the target/culprit or non-target/non-culprit lesion (nanosecond) | 6 month
  6-month changes in healed phenotype FLIm measurement
6-month temporal changes in FLIm measurement of plaque calcification in the target/culprit or non-target/non-culprit lesion (nanosecond) | 6 month
  6-month changes in calcification FLIm measurement

CONTACTS AND LOCATIONS:
Overall Officials: Sunwon Kim, MD, PhD, Study Director — Korea University Ansan Hospital; Dong Oh Kang, MD, PhD, Study Director — Korea University Guro Hospital; Jin Won Kim, MD, PhD, Principal Investigator — Korea University Guro Hospital; Hongki Yoo, PhD, Study Director — Korea Advanced Institute of Science and Technology
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee MW, Song JW, Kang WJ, Nam HS, Kim TS, Kim S, Oh WY, Kim JW, Yoo H. Comprehensive intravascular imaging of atherosclerotic plaque in vivo using optical coherence tomography and fluorescence lifetime imaging. Sci Rep. 2018 Sep 28;8(1):14561. doi: 10.1038/s41598-018-32951-9. PMID 30267024
- [Background] Kim S, Yoo H, Kim JW. Long Journey of Intravascular Imaging: What and How to Look at the Atheroma in Coronary Artery. JACC Cardiovasc Imaging. 2021 Sep;14(9):1843-1845. doi: 10.1016/j.jcmg.2020.11.015. Epub 2020 Dec 16. No abstract available. PMID 33341412
- [Background] Nam HS, Kang WJ, Lee MW, Song JW, Kim JW, Oh WY, Yoo H. Multispectral analog-mean-delay fluorescence lifetime imaging combined with optical coherence tomography. Biomed Opt Express. 2018 Mar 27;9(4):1930-1947. doi: 10.1364/BOE.9.001930. eCollection 2018 Apr 1. PMID 29675330